CLINICAL TRIAL: NCT04447131
Title: Effect of SARS-CoV-2 Infection on Platelet Aggregation and Other Coagulation Parameters
Brief Title: Effect of COVID-19 on Platelet Aggregation
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Director of Coronary Care Unit, University of Sao Paulo
Other Study IDs: SDC 5089/20/118
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: Platelet aggreggation; COVID-19; SARS-CoV-2; Multiplate
MeSH Terms: conditions — COVID-19 | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19: Confirmation of the diagnosis of COVID-19 by laboratory method (RT-PCR and / or positive serology for SARS-CoV-2 - COVID group).
  Interventions: Other: venipuncture in peripheral vein
- Healthy Individuals: Asymptomatic and with negative SARS-CoV-2 serology
  Interventions: Other: venipuncture in peripheral vein
- Respiratory symptoms but negative for COVID-19: Negative for SARS-CoV-2. But with respiratory symptoms
  Interventions: Other: venipuncture in peripheral vein

INTERVENTIONS:
Other: venipuncture in peripheral vein — single vacuum venipuncture in peripheral vein

SUMMARY:
This is a mechanistic, observational, prospective, case and control study, to compare platelet aggregation, analyzed by Multiplate-ADP, in hospitalized patients diagnosed with COVID-19 versus healthy controls. Thus will be included 60 patients who present with respiratory symptoms within 72 hours of hospitalization and confirmation of the diagnosis of COVID-19 by laboratory method (RT -PCR and / or positive serology for SARS-CoV-2 - COVID group); this group will be compared to 60 healthy individuals (asymptomatic and with negative SARS-CoV-2 serology), matched by sex and age to the previous group.

DETAILED DESCRIPTION:
There is strong evidence that SARS-CoV-2 infection is associated with atherothrombotic phenomena. However, platelet activity in COVID-19 has not yet been studied.

Thus, the main objective of this project is to evaluate platelet aggregation by the Multiplate-ADP method in hospitalized patients diagnosed with COVID-19, in comparison with the platelet aggregation evaluated by the same method in healthy controls.

Secondary objectives include the assessment of parameters related to coagulation, inflammation, and clinical outcome variables.

This is a mechanistic, observational, prospective, case and control study, which will include 60 patients who present with respiratory symptoms within 72 hours of hospitalization and confirmation of the diagnosis of COVID-19 by laboratory method (RT -PCR and / or positive serology for SARS-CoV-2 - COVID group); this group will be compared to 60 healthy individuals (asymptomatic and with negative SARS-CoV-2 serology), matched by sex and age to the previous group.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to sign the Free and Informed Consent Form (ICF).
* Case group: patients with up to 72 hours of hospitalization for respiratory symptoms.
* Control group: healthy volunteers, defined as having no history (confirmed or suspected) of COVID-19 or chronic diseases (except hypertension, obesity, dyslipidemia)

Exclusion Criteria:

* Known platelet dysfunction or platelet count <100,000 / µL or> 450,000 / µL;
* Terminal illness;
* Known liver disease or clotting disorder;
* Hematocrit less than 34% or greater than 55%;
* Previous use of antiplatelet agents and / or anticoagulants (except acetylsalicylic acid and prophylactic heparin);
* Patients on invasive mechanical ventilation or receiving high oxygen flow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with up to 72 hours of hospitalization for respiratory symptoms, tested with RT- PCR for respiratory viruses, will be evaluated for inclusion. Patients with diagnostic criteria for COVID-19 will be considered a case group (COVID-19 group) and will be compared to two other groups: patients hospitalized for respiratory symptoms with a negative test for SARS-CoV-2, and healthy control group.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation analyzed by Multiplate-ADP | at inclusion
  Compare platelet aggregation analyzed by Multiplate-ADP in hospitalized patients diagnosed with COVID-19 versus healthy controls.

SECONDARY OUTCOMES:
Platelet aggregation by Multiplate-ASPI and Multiplate-TRAP in patients hospitalized for COVID-19 versus healthy controls. | at inclusion
  Compare platelet aggregation by Multiplate-ASPI and Multiplate-TRAP in patients hospitalized for COVID-19 versus healthy controls.
Reticulated platelet fraction in patients hospitalized for COVID-19 versus healthy controls. | at inclusion
  Compare the levels of the reticulated platelet fraction in patients hospitalized for COVID-19 versus healthy controls.
Platelet aggregation for COVID-19 versus patients hospitalized for respiratory symptoms but negative for COVID-19. | at inclusion,
  Compare platelet aggregation by Multiplate-ADPMultiplate-ASPI and Multiplate-TRAP in patients hospitalized for COVID-19 versus patients hospitalized for respiratory symptoms but negative for COVID-19.
Reticulated platelet fraction in patients hospitalized for COVID-19 versus patients hospitalized for respiratory symptoms but negative for COVID-19 research. | at inclusion
  Compare the levels of the reticulated platelet fraction in patients hospitalized for COVID-19 versus patients hospitalized for respiratory symptoms but negative for COVID-19.
Platelet aggregation in patients hospitalized for COVID-19 versus patients hospitalized for Influenza. | at inclusion
  Compare platelet aggregation by Multiplate-ADP, Multiplate-ASPI and Multiplate-TRAP in patients hospitalized for COVID-19 versus patients hospitalized for Influenza.
Reticulated platelet fraction in patients hospitalized for COVID-19 versus patients hospitalized for Influenza. | at inclusion
  Compare the levels of the reticulated platelet fraction in patients hospitalized for COVID-19 versus patients hospitalized for Influenza.
Platelete aggreggation versus composite outcome of death from any cause, thrombotic events, need for ICU, need for intubation during hospitalization | at inclusion
  Compare the levels of platelet aggregation (by Multiplate ADP, ASPI and TRAP) in patients with or without the composite outcome of death from any cause, thrombotic events, need for ICU, need for intubation during hospitalization Compare the levels of platelet aggregation (by Multiplate ADP, ASPI and TRAP) in patients with or without the composite outcome of death from any cause, thrombotic events, need for ICU, need for intubation during hospitalization
Reticulated platelet fraction versus composite outcome of death from any cause, thrombotic events, need for ICU, need for intubation during hospitalization | at inclusion
  Compare the levels of the reticulated platelet fraction in patients with or without the composite outcome of death from any cause, thrombotic events, need for ICU, need for intubation during hospitalization;
Platelet aggregation versus time (days) of total hospitalization and in the ICU | at inclusion
  Compare the levels of platelet aggregation (by Multiplate ADP, ASPI and TRAP) with the time (days) of total hospitalization and in the ICU;
Reticulated platelet fraction versus time (days) of total hospitalization and in the ICU | at inclusion
  Correlate the levels of the reticulated platelet fraction with the time (days) of total hospitalization and in the ICU;

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Instituto do Coracao (InCor), Hospital das Clinicas HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo
  - Instituto de infectologia Emílio Ribas, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwong JC, Schwartz KL, Campitelli MA, Chung H, Crowcroft NS, Karnauchow T, Katz K, Ko DT, McGeer AJ, McNally D, Richardson DC, Rosella LC, Simor A, Smieja M, Zahariadis G, Gubbay JB. Acute Myocardial Infarction after Laboratory-Confirmed Influenza Infection. N Engl J Med. 2018 Jan 25;378(4):345-353. doi: 10.1056/NEJMoa1702090. PMID 29365305
- [Background] Hottz ED, Bozza FA, Bozza PT. Platelets in Immune Response to Virus and Immunopathology of Viral Infections. Front Med (Lausanne). 2018 Apr 30;5:121. doi: 10.3389/fmed.2018.00121. eCollection 2018. PMID 29761104
- [Background] McNicol A, Israels SJ. Beyond hemostasis: the role of platelets in inflammation, malignancy and infection. Cardiovasc Hematol Disord Drug Targets. 2008 Jun;8(2):99-117. doi: 10.2174/187152908784533739. PMID 18537597
- [Background] Corrales-Medina VF, Madjid M, Musher DM. Role of acute infection in triggering acute coronary syndromes. Lancet Infect Dis. 2010 Feb;10(2):83-92. doi: 10.1016/S1473-3099(09)70331-7. PMID 20113977
- [Background] Rondina MT, Brewster B, Grissom CK, Zimmerman GA, Kastendieck DH, Harris ES, Weyrich AS. In vivo platelet activation in critically ill patients with primary 2009 influenza A(H1N1). Chest. 2012 Jun;141(6):1490-1495. doi: 10.1378/chest.11-2860. Epub 2012 Mar 1. PMID 22383669
- [Background] Le VB, Schneider JG, Boergeling Y, Berri F, Ducatez M, Guerin JL, Adrian I, Errazuriz-Cerda E, Frasquilho S, Antunes L, Lina B, Bordet JC, Jandrot-Perrus M, Ludwig S, Riteau B. Platelet activation and aggregation promote lung inflammation and influenza virus pathogenesis. Am J Respir Crit Care Med. 2015 Apr 1;191(7):804-19. doi: 10.1164/rccm.201406-1031OC. PMID 25664391
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Rubak P, Villadsen K, Hvas AM. Reference intervals for platelet aggregation assessed by multiple electrode platelet aggregometry. Thromb Res. 2012 Sep;130(3):420-3. doi: 10.1016/j.thromres.2012.06.017. Epub 2012 Jul 17. PMID 22809844
- [Derived] Bertolin AJ, Dalcoquio TF, Salsoso R, de M Furtado RH, Kalil-Filho R, Hajjar LA, Siciliano RF, Kallas EG, Baracioli LM, Lima FG, Giraldez RR, Cavalheiro-Filho C, Vieira A, Strunz CMC, Giugliano RP, Tantry US, Gurbel PA, Nicolau JC. Platelet Reactivity and Coagulation Markers in Patients with COVID-19. Adv Ther. 2021 Jul;38(7):3911-3923. doi: 10.1007/s12325-021-01803-w. Epub 2021 Jun 4. PMID 34086266